CLINICAL TRIAL: NCT06894290
Title: International Cardiac Amyloidosis Registry
Acronym: ICAR
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Nina Ajmone Marsan, MD, PhD, Leiden University Medical Center
Other Study IDs: ICAR
Record Dates: First submitted 2025-03-12; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Amyloidosis
Keywords: Cardiac amyloidosis; ATTR amyloidosis; AL amyloidosis; Echocardiography
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CA: Patients diagnosed with cardiac amyloidosis. Either ATTR-CA or AL-CA.

SUMMARY:
Cardiac amyloidosis is a relatively rare disease. However, with the newer imaging techniques that have become available to us in recent years, determining the diagnosis is becoming more common. There are several variants. Each variant involves protein accumulation between heart muscle cells. This leads to the heart stiffening and, as a result, the heart has a hard time filling. This can lead to heart failure with complaints such as fluid retention, cardiac arrhythmias such as atrial fibrillation, conduction abnormalities that sometimes require a pacemaker, and clot formation in the heart that can cause a stroke and narrowing of the aortic valve. Getting the correct diagnosis is important because specific treatment is available in some cases for the different variants of cardiac amyloidosis. This research is needed to better understand the course of this disease profile and which patients respond well to the specific treatment.

The aim of this research is to find out more about the course of the cardiac amyloidosis disease. The investigators see to what extent patients deteriorate in their condition due to the disease and how often they need to be hospitalized. Furthermore, the investigators want to learn to what extent certain abnormalities (on e.g. cardiac ultrasound) can predict how quickly clinical deterioration occurs. Finally, for certain forms of cardiac amyloidosis there is a specific drug treatment. Through this research, the investigators want to try to determine who really benefits from the specific medication in order to prescribe it to the right patients.

DETAILED DESCRIPTION:
Rationale: Patients with cardiac amyloidosis are in general underdiagnosed and undertreated. AL amyloidosis is a disease with a very poor prognosis if left untreated. For ATTR amyloidosis, recently, specific treatment has become available for patients fulfilling certain criteria with good results in clinical trials. The rationale behind this prospective registry is to collect real-world data on diagnostic process, management, progression of disease and outcome of patients with cardiac AL and ATTR amyloidosis who are treated following local standards and to obtain (echocardiographic) predictors of prognosis in these patients.

Objective: The objective of the study is to evaluate the diagnostic process from onset symptoms to diagnosis, the outcome in a real-world cohort of amyloidosis patients and to find predictors (both clinical and echocardiographic) of outcome Study design: Prospective long-term observational study Study population: All patients >18 years old, prospectively diagnosed with cardiac AL or ATTR amyloidosis Intervention (if applicable): n/a Main study parameters/endpoints: The main study endpoints are death, heart failure hospitalization and cardiovascular events Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients who participate in the registry will undergo structured follow up according to the clinical care pathway for amyloidosis patients based on the recommendations in the most recent Position Statement from the European Society of Cardiology [1]. There will be no additional visits planned, therefore no additional burden is associated with participation in the registry. Patients agree that their anonymized data is shared with other centers within the amyloidosis consortium.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with AL or ATTR cardiac amyloidosis following the recommendations of the European Society of Cardiology [1] which include:

Signs and symptoms, ECG, echo or CMR suggestive of cardiac amyloidosis and

* negative hematological test and bone scintigraphy Perugini stage 2 or 3 (is diagnostic for ATTR amyloidosis)
* negative hematological test and bone scintigraphy Perugini stage 1 and histological confirmation (either extracardiac or cardiac biopsy) with subtyping of ATTR amyloidosis
* positive hematological test and bone scintigraphy Perugini stage 1-3 and histological confirmation (usually cardiac biopsy) with subtyping of ATTR amyloidosis
* positive hematological rest and bone scintigraphy Perugini stage 0, MRI consistent with amyloidosis and histological confirmation (either extracardiac or cardiac biopsy) with subtyping AL amyloidosis

Exclusion Criteria:

* Unable to provide informed consent due to insufficient language proficiency or intellectual capabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with diagnosis of AL or ATTR diagnosis will be prospectively included from 1st of January 2023 in the registry (if consent is provided). Currently, about 10 patients per year are diagnosed in the LUMC, therefore multicenter cooperation is needed to include sufficient patients. We have a consortium of at least 15 centers that are willing to participate. Therefore we estimate an inclusion of ~150 patients per year. The rate of diagnosis will probably increase with increasing awareness for amyloidosis, with potentially increasing inclusion rates. An estimated 1/3 of patient will have AL and 2/3 will have ATTR amyloidosis.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1 year
  The main study endpoint is all-cause mortality

SECONDARY OUTCOMES:
Progression | 1 year
  Progression of disease (defined by disease specific progression stages such as Mayo score for AL amyloidosis and NAC score for ATTR amyloidosis)
HFH | 1 year
  Heart failure hospitalization
Events | 1 year
  Cardiovascular events (including cerebrovascular accident and other thromboembolic events, cardiac arrhythmias and pacemaker implantations)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Ajmone Marsan, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (6):
- Belgium (2):
  - AZ St Jan, Bruges
  - UZ Antwerpen, Edegem
- Fondazione Policlinico Universitario 'A. Gemelli' IRCCS, Roma, Roma, Italy
- Kitasato University Hospital, Sagamihara, Japan
- Leiden University Medical Center, Leiden, Netherlands
- Santa Marta Hospital, CHULC, Lisbon, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No
We will share individual participant data between centers when asked for, but we will not make it public available

REFERENCES:
- [Background] Bukhari S, Khan SZ, Bashir Z. Atrial Fibrillation, Thromboembolic Risk, and Anticoagulation in Cardiac Amyloidosis: A Review. J Card Fail. 2023 Jan;29(1):76-86. doi: 10.1016/j.cardfail.2022.08.008. Epub 2022 Sep 17. PMID 36122817
- [Background] Maurer MS, Schwartz JH, Gundapaneni B, Elliott PM, Merlini G, Waddington-Cruz M, Kristen AV, Grogan M, Witteles R, Damy T, Drachman BM, Shah SJ, Hanna M, Judge DP, Barsdorf AI, Huber P, Patterson TA, Riley S, Schumacher J, Stewart M, Sultan MB, Rapezzi C; ATTR-ACT Study Investigators. Tafamidis Treatment for Patients with Transthyretin Amyloid Cardiomyopathy. N Engl J Med. 2018 Sep 13;379(11):1007-1016. doi: 10.1056/NEJMoa1805689. Epub 2018 Aug 27. PMID 30145929
- [Background] Garcia-Pavia P, Rapezzi C, Adler Y, Arad M, Basso C, Brucato A, Burazor I, Caforio ALP, Damy T, Eriksson U, Fontana M, Gillmore JD, Gonzalez-Lopez E, Grogan M, Heymans S, Imazio M, Kindermann I, Kristen AV, Maurer MS, Merlini G, Pantazis A, Pankuweit S, Rigopoulos AG, Linhart A. Diagnosis and treatment of cardiac amyloidosis. A position statement of the European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Eur J Heart Fail. 2021 Apr;23(4):512-526. doi: 10.1002/ejhf.2140. Epub 2021 Apr 7. PMID 33826207